CLINICAL TRIAL: NCT02592031
Title: An Open, Randomized, Two-way Cross-over Phase I Study to Compare the Bioavailability, Safety and Tolerability of Single s.c. Doses of 300 IU XM17 With 300 IU Gonal-f® in 36 Healthy, Down-regulated Young Women
Brief Title: Study to Compare the Bioavailability, Safety and Tolerability of XM17 in Healthy, Down Regulated Young Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merckle GmbH (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XM17-02; 2008-005756-24 (EudraCT Number)
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Bioequivalence
MeSH Terms: interventions — follitropin alfa; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- XM17 (Experimental): XM17 will be administered by 1 mL syringes in graduated steps of 0.01 mL.
  Interventions: Drug: XM17
- Gonal-f® (Experimental): Gonal-f® will be provided in pens with integrated vials of 0.5 mL
  Interventions: Drug: Gonal-f®
- Zoladex® (Active Comparator): Zoladex® 3.6 mg will be administered by subcutaneous injection
  Interventions: Drug: Zoladex®

INTERVENTIONS:
Drug: XM17 — 300 IU corresponds to an injection volume of 0.5 mL.
  Arms: XM17
Drug: Gonal-f® — 300 IU corresponds to an injection volume of 0.5 mL.
  Other Names: follitropin alfa
  Arms: Gonal-f®
Drug: Zoladex® — 3.6 mg
  Other Names: goserelin acetate
  Arms: Zoladex®

SUMMARY:
Aim of this study is to demonstrate the bioequivalence of single subcutaneous doses of XM17 and Gonal-f® in a confirmatory design. Furthermore, safety and tolerability will be assessed in human healthy female subjects. Only female subjects will be included in the study to reach the objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

* Having signed written informed consent
* Healthy female subjects of any racial origin
* 18-39 years at the time of screening
* Body mass index (BMI) between 18-29 kg/m2 and a body weight of ≥ 50 kg
* Use of oral contraceptives for contraceptive purposes only and not for regularization of menstrual cycle, for at least 3 months
* Normal uterus and two functioning ovaries
* Agrees to use an adequate method of contraception during the study
* Non-smoking or moderate smokers of < 10 cigarettes a day

Exclusion Criteria:

* Pregnancy
* Polycystic ovary syndrome, impaired ovarian function, severe endometriosis class III or IV, submucosal myoma uteri
* History of endocrine abnormalities with treatment within the last six months.
* Contraindications for the use of gonadotropins and goserelin
* Breast-feeding or being within a period of 2 months after delivery or abortion.
* Use of an injectable hormonal contraceptive within a period of 6 months prior to screening
* Treatment in the previous three months with any drug known to have a well-defined potential for toxicity to a major organ

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Comparison of single dose pharmacokinetics (Cmax) | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  XM17 and Gonal-f® tested statistically for bioequivalence.
Comparison of single dose pharmacokinetics (AUC0-t) | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  XM17 and Gonal-f® tested statistically for bioequivalence.

SECONDARY OUTCOMES:
Pharmacokinetics AUC0-∞ | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Area under the XM17 / Gonal-f® concentration time curve from time 0 extrapolated to infinity
Pharmacokinetics AUC0-168h | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Area under the XM17 / Gonal-f® concentration time curve from time 0 to 168 h
Pharmacokinetics Cmax,obs | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Maximum XM17 / Gonal-f® concentration determined during the interval of sample taking
Pharmacokinetics Tmax | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Time to maximum XM17 / Gonal-f® concentration
Pharmacokinetics λZ | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Apparent terminal elimination rate constant.
Pharmacokinetics t1/2 | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Apparent terminal elimination half life.
Pharmacokinetics CL/F | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Serum clearance after dosing
Pharmacokinetics Vz/F | Pre-dose at -10 min, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Volume of Distribution during the terminal phase after extravascular administration
Percentage of participants with adverse events | Signing of informed consent to final data collection (27 days)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.

REFERENCES:
- [Derived] Lammerich A, Mueller A, Bias P. Phase I, two-way, crossover study to demonstrate bioequivalence and to compare safety and tolerability of single-dose XM17 vs Gonal-f(R) in healthy women after follicle-stimulating hormone downregulation. Reprod Biol Endocrinol. 2015 Dec 1;13:130. doi: 10.1186/s12958-015-0124-y. PMID 26621118